CLINICAL TRIAL: NCT00309426
Title: The Effect of Serum Fetuin A Concentration on the 5-Year Prognosis in Hemodialysis Patients
Brief Title: Effect of Fetuin A in Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Shizuoka (Other)
Collaborators: Maruyama Memorial General Hospital (Other)
Other Study IDs: CT2006003
Record Dates: First submitted 2006-03-27; First posted 2006-03-31 (Estimated); Last update posted 2006-05-22 (Estimated); Status verified 2006-03

CONDITIONS: Hemodialysis; Malnutrition
Keywords: atherosclerosis
MeSH Terms: conditions — Malnutrition; Atherosclerosis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of this study is to examined the effect of fetuin A on atherosclerosis and prognosis in hemodialysis patients.

DETAILED DESCRIPTION:
Fetuin A is known to be a potent inhibitor of ectopic calcification in plasma, and the concentration of fetuin A is closely associated with protein nutritional status. The purpose of this study is to examine whether the plasma concentration of fetuin A is associated with atherosclerosis and 5-year prognosis in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis for at least 6 months

Exclusion Criteria:

* Disabled patients

Ages: 0 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 2001-03; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: Hiromichi Kumagai, MD, Study Chair — University of Shizuoka
Locations (1):
- Maruyama Hospital, Hamamatsu, Shizuoka, Japan